CLINICAL TRIAL: NCT06300034
Title: Parental Perceptions and Acceptance of Silver Diamine Fluoride Staining in Italy: A Cross-sectional Study
Brief Title: Parental Perceptions and Acceptance of Silver Diamine Fluoride in Italy
Acronym: SDF
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Simone Bagattoni, Principal investigator, University of Bologna
Other Study IDs: bagattoni2
Record Dates: First submitted 2024-02-23; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Perceptions; Acceptability; SDF
Keywords: Silver Diamine Fluoride; Parental perceptions and acceptance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
Parental perceptions on staining due to Silver Diamine Fluoride (SDF) could affect its implementation in pediatric dentistry. This study represents the second part of a wider project focused on SDF aesthetic acceptability among Italian parents.

DETAILED DESCRIPTION:
The aim of this survey was to assess the parental acceptance of Silver Diamine Fluoride (SDF) staining in Italy, and to examine wether the level of acceptability depends on location, child's behavior, or demographic background. A cross-sectional study was undertaken, involving 234 Italian parents whose children were attending two university dental clinics. Using a validated Italian version of the questionnaire 'Parental Perceptions of Silver Diamine Fluoride Dental Color Changes', researchers administered a series of closed-ended Likert-type questions to parents. The questionnaire included sets of colored photographs showing both anterior and posterior teeth before and after SDF treatment. Respondents were requested to provide their assessments based on the presented visual stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Italian-speaking parents
* Parents of healthy children or children with mild systemic disease. American Society of Anesthesiologists (ASA) status 1-2
* Parents of children under the age of 12 years
* Parents of children with previous caries experience in primary teeth
* Parents who consented to participate

Exclusion Criteria:

* No Italian-speaking parents
* Parents of children with ASA status ≥ 3
* Parents of children over the age of 12 years
* Parents of children without previous caries experience in primary teeth
* Parents who no consented to participate

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Parents awaiting their child's dental appointments at two distinct locations: the Unit of Dental Care for Special Needs Patients and Paediatric Dentistry at the University of Bologna, Bologna, Italy, and the Unit of Paediatric Dentistry at the University of Pisa, Pisa, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Parental overall acceptance of SDF staining on anterior and posterior teeth | Baseline
  Measurement tool: questionnaire. Specific questions focused on the general acceptability of the visible SDF staining for anterior and posterior teeth. Scores for levels of acceptability were 'unacceptable' (scoring 1), 'somewhat unacceptable' (scoring 2), 'somewhat acceptable' (scoring 3), and 'acceptable' (scoring 4). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Parental willingness to accept SDF treatment on anterior and posterior teeth depending on child's behavior | Baseline
  Measurement tool: questionnaire. Acceptance of SDF treatment was evaluated by asking parents if they would allow the treatment to be done on their children in a context of hypothetical scenarios of child cooperation (child cooperative; child upset but could cooperate; child crying; child needs physical restraint; child screaming or kicking; child needs nitrous oxide sedation; child needs oral sedation; child needs general anesthesia). This assessment was carried out separately for anterior and posterior teeth. Scores for acceptance level were 'extremely unlikely' (scoring 1), 'somewhat unlikely' (scoring 2), 'somewhat likely' (scoring 3), and 'very likely' (scoring 4). Higher scores mean a better outcome.
Parental overall acceptability of SDF staining according to demographic background | Baseline
  Measurement tool: questionnaire. Specific questions were strategically formulated to capture a comprehensive range of demographic variables of the participants, including factors such as age, education, and socioeconomic status. The findings from this analysis contribute valuable insights into the nuanced relationship between demographic characteristics and parental attitudes towards SDF staining in the Italian context.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Bagattoni, Principal Investigator — Bologna University
Locations (1):
- Servizio di Assistenza Odontoiatrica per disabili in età evolutiva e di odontoiatria infantile, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No